CLINICAL TRIAL: NCT04708002
Title: How to Improve the Care of Elderly People From Nursing Home: Interventional Research With Mixed Methods on an Early Integrated Palliative Approach
Brief Title: Interventional Research With Mixed Methods on an Early Integrated Palliative Approach in Nursing Home
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maison Médicale Jeanne Garnier (Other)
Collaborators: Ministry of Health, France (Other Government); Regional Agency for Health PACA (Other); Groupement Interrégional de Recherche Clinique et d'Innovation (Other); Versailles Saint-Quentin-en-Yvelines University (Other); Centre hospitalier de l'Université de Montréal (CHUM) (Other); École de santé publique Université de Montréal (Unknown); Centre Hospitalier Henri Duffaut - Avignon (Other); Maison de santé Marie Galène (Unknown); Agence Regionale de Sante d'Ile de France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020-A01832-37
Record Dates: First submitted 2020-12-03; First posted 2021-01-13 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-01

CONDITIONS: Palliative Care; Nursing Homes; Aged
Keywords: Integrated and early palliative care approach; care pathway; quality of care; intervention research; resident; nursing home caregiver; health services research; mixed method

STUDY DESIGN:
Intervention Model Description: stepped-wedge design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- First EIPCA-NH group (Other): There are 5 nursing home in each arm (cluster), randomly selected from 3 French areas.
  Interventions: Other: early integrated palliative approach model
- Early intermediate EIPCA-NH group (Other): There are 5 nursing home in each arm (cluster), randomly selected from 3 French areas.
  Interventions: Other: early integrated palliative approach model
- Late intermediate EIPCA-NH group (Other): There are 5 nursing home in each arm (cluster), randomly selected from 3 French areas.
  Interventions: Other: early integrated palliative approach model
- Last EIPCA-NH group (Other): There are 5 nursing home in each arm (cluster), randomly selected from 3 French areas.
  Interventions: Other: early integrated palliative approach model

INTERVENTIONS:
Other: early integrated palliative approach model — From the construction of a common vision of palliative care between actors inside and outside the nursing home to the sustainability of palliative care in nursing home.

SUMMARY:
The national context of the end of life of elderly people living in Nursing Home (NH) is concerning.

A quarter of NH residents die each year representing a quarter of annual deaths in France of all ages. The number of resident deaths arises (148,300 deaths in 2015 versus 124,500 in 2011). In fact, the age of residents welcomed in NH increase, 82% of residents are 80 years old and over, suffering from several chronic pathologies, some of which are serious and incurable. These are the main cause of death for residents. The advancing age of NH residents and the interweaving of multiple chronic conditions and disabling pathologies generate complex care needs, the complexity of which undermines the current system of care organization. In 2016, 59% of NH residents were severely dependent in their activities of daily living (ADL) and instrumental activities of daily living (IADL) according to the French scale Autonomie, Gérontologie Groupe Iso Ressources, (1 the most dependant to 6 the less dependent); the majority of these most dependent NH residents (80% of Groupe Iso-Ressource 1-2 in 2011) had at least one unstable chronic pathology and 73% of deceased residents (in 2015) come from this group whose level of dependence is very high.

Palliative care (PC), which is care focused on maintaining quality of life in a context of incurable and complex pathology, therefore appears to be indicated in the context of NH. However, residents' access to PC remains limited, uneven and late. The number of residents requiring this support is estimated at more than 100,000 residents per year. The consequences of such situation are serious, first with regard to the quality of life of NH residents and their family caregivers, but also the inappropriate use of health services (as shown by the excessive use of emergency department and unscheduled hospitalizations) and work life for care providers in NH is affected (care providers suffer from a lack of support when faced with the difficulties of caring for NH residents at the end of their life). However, these consequences are potentially avoidable by means of adapted organizational solutions. The implementation of an integrated and early palliative approach (IEPA) in care pathway of patient is one of the solutions recommended by the World Health Organization and the French National Authority for Health. Several studies have shown the benefit of such approach in the management of cancer patients. However, the transferability and effectiveness of this approach in other organizational and population contexts are poorly documented, particularly in NH settings.

The main objective is to evaluate, through a pragmatic controlled trial the effectiveness of an Early Integrated Palliative Care Approach in usual NH context (EIPCA-NH) on the quality of care in NH for elderly in need of PC. The secondary objectives concern:

1. the implementation process of the EIPCA-NH: i) measure the degree of implementation of the EIPCA-NH in each site, ii) identify and understand the factors (individual and organizational) facilitating or limiting the success of the implementation process of an IEPA according to NH contexts (inter-site comparison).
2. the effects of the EIPCA-NH in the NH : i) on the quality of life of residents requiring PC and ii) that of their family caregivers, iii) on the quality work life of professional caregivers and iv) on the care pathway of NH residents.

A mixed methods research, with qualitative and quantitative approach, will be carried out in at least 20 NH in three different health territories. These NH will benefit from a EIPCA-NH intervention which consists of 1) implementing a mechanism for sharing and co-producing knowledge, 2) integrating this approach as early as possible in the care of residents. This study is based on a multicenter, randomized crossover cluster-type stepped-wedge study, running on 4 years in order to measure the sustainability of EIPCA-NH; the quantitative analysis of the effectiveness of EIPCA-NH will focus on an open cohort of 3,500 residents receiving the intervention. The qualitative component will consist of a multiple case study to analyse the process of implementation and production of the EIPCA-NH. The integrative analysis of qualitative and quantitative data will allow a better understanding of the causal mechanisms of the observed phenomena.

This project will provide evidence on the value of EIPCA and the conditions for its implementation and transferability. The proposed intervention will help improve care practices for all NH residents (600,000 people). The approach by co-construction between actors of the thousands of care structures (NH, cities, hospitals) and researchers should promote a better representation of PC, promote the culture of anticipation, evaluation and collaboration between actors of in- and out- NH, contributing to a better synergy of intersectoral and territorial actions of the supply of health services.

ELIGIBILITY:
Inclusion Criteria:

* Be a resident of a nursing home.
* Be 60 years of age or older.
* Be a resident who has been identified by the Proactive identification Guidance

Exclusion Criteria:

* Be under 60 years of age.
* Resident living temporarily in the nursing home.
* Refusing to participate

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3500 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in the number of resident with access to palliative care assessed by the proactive identification guidance and by the InterRAI Palliative Care assessment system | Quantitative data will be collected throughout study completion (up to 2 years), each nursing home will have evaluations following a stepped-wedge design with 4 time periods: Pre-implantation, Implantation, Post implantation, Sustainability
  stepped-wedge with 4 clusters

SECONDARY OUTCOMES:
Median score of the degree of implementation using a scale based on Proctor et al indicators, with a minimum score of 6 and a maximum score of 30. | Qualitative data collections will be carry out continuously throughout study completion (up to 2 years)
  stepped-wedge with 4 clusters : The minimum score is 6 which means that the degree of implementation is very low. The maximum score is 30 which means that the degree of implementation is very high.
Median score of quality of life of nursing home resident using InterRAI Self-Report Nursing Home Quality of Life Survey instrument (interRAI-QoL) | Quantitative data collections will be done throughout study completion (up to 2 years), each nursing home will have one evaluation following a stepped-wedge design with 2 time periods: Pre-implantation, Post implantation
  stepped-wedge with 4 clusters : InterRAI quality of life has ten subscales with minimum score of 0 and a maximum score ranging between 16 to 24. The minimum score (0) is the best outcome for quality of life and, the maximum (16-24) is the worse outcome.
Median score of quality of life of informal caregiver using the Caregiver's Burden Scale in End-of-Life Care (CBS-EOLC) self-questionnaire | Quantitative data collections will be done throughout study completion (up to 2 years), each nursing home will have one evaluation following a stepped-wedge design with 2 time periods: Pre-implantation, Post implantation
  stepped-wedge with 4 clusters : The minimum score is 16 meaning that it is the best outcome for the quality of life of informal caregivers and, the maximum score is 54 meaning that it is the worst outcome.
Median score of quality of life of professional caregiver using the professional quality of life scale (ProQoL) | Quantitative data collections will be done throughout study completion (up to 2 years), each nursing home will have one evaluation following a stepped-wedge design with 2 time periods: Pre-implantation, Post implantation
  stepped-wedge with 4 clusters : The minimum score is 30, the average score is around 50 and the highest score is 57 or over. The highest score means a good quality of life of professional caregiver and the lowest score means a poor professional caregiver's quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Bagaragaza, MPH, PhD, Principal Investigator — SPES, Maison médicale Jeanne Garnier; Frédéric Guirimand, MD, PhD, Principal Investigator — SPES, Maison médicale Jeanne Garnier; Philippe Aegerter, MD, PhD, Principal Investigator — GIRCI IDF
Locations (3):
- France (3):
  - Ch Avignon, Avignon
  - Maison de Santé Marie Galène, Bordeaux
  - Maison Médicale Jeanne Garnier, Paris

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: Study protocole: july 2021

REFERENCES:
- [Derived] Umubyeyi B, Leboul D, Bagaragaza E. "You close the door, wipe your sadness and put on a smiling face": a qualitative study of the emotional labour of healthcare professionals providing palliative care in nursing homes in France. BMC Health Serv Res. 2024 Sep 16;24(1):1070. doi: 10.1186/s12913-024-11550-7. PMID 39278920
- [Derived] Bagaragaza E, Colombet I, Perineau M, Aegerter P, Guirimand F. Assessing the implementation and effectiveness of early integrated palliative care in long-term care facilities in France: an interventional mixed-methods study protocol. BMC Palliat Care. 2023 Apr 6;22(1):35. doi: 10.1186/s12904-023-01157-w. PMID 37024830